CLINICAL TRIAL: NCT01629628
Title: An Investigator Initiated Prospective, Single Center, Randomized, Open Label Study to Assess the Efficacy of Adalimumab for the Maintenance of Remission in Post-operative CD Patients
Brief Title: Adalimumab for the Management of Post-operative Crohn's Disease (CD)
Acronym: POPART
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, director, R&D Division, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-10-ES-0446-TLV-CTIL
Record Dates: First submitted 2012-06-19; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Colitis Granulomatous; Crohn's Disease; Enteritis Regional; Ileitis Regional; Ileitis Terminal; Ileocolitis
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab; Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab (Experimental)
  Interventions: Drug: Adalimumab
- 6-mercaptopurine (Active Comparator)
  Interventions: Drug: 6 Mercaptopurine

INTERVENTIONS:
Drug: Adalimumab — Subcutaneous adalimumab injections, loading dose of 160 mg and 80 mg on 0 and 2 weeks and maintenance of 40 mg every other week for the duration of the study.
  Other Names: Humira
  Arms: Adalimumab
Drug: 6 Mercaptopurine — 6MP will be administered orally starting at a dose of 6MP of 50mg/day with escalating doses every 1-2 weeks as tolerated, to a target dose of 1-1.5 mg/kg.
  --------------------------------------------------------------------------------
  Other Names: Purinethol
  Arms: 6-mercaptopurine

SUMMARY:
This study will be a prospective, open label, randomized, comparative study. Comparing the efficacy of adalimumab with immunomodulator therapy (i.e. 6-mercaptopurine, 6-MP), in maintaining remission of post-operative CD patients, with a high risk of disease recurrence.

Patient assessment for efficacy will be conducted through interval endoscopic surveillance at 24 and 52 weeks.

Patients in the adalimumab arm, showing endoscopic remission at 52 weeks of therapy, will be re-randomized to either maintain adalimumab therapy for an additional 52 weeks or conclude therapy. A third endoscopic assessment for these patients will be conducted at 104 weeks.

The investigators expect a substantial increase in both endoscopic, as well as clinical remission rate in patients on adalimumab therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old at the time of screening
* Male or female
* Firs ileocolonic surgical resection (
* Evidence of both macroscopic as well an microscopic evidence of Crohn's disease in the resected intestinal segment
* Patient able to undergo pre randomization screening no earlier then 14 days and no later then 45 days post operatively.
* Patients may receive anti-TNF-agents (i.g. infliximab or adalimumab)previously
* Patients may receive corticosteroids, 6MP/AZA, methotrexate, or mesalamine prior to surgery.
* Antibiotics, or mesalamine, must be discontinued within the screening/baseline 4 week period. Patients on steroids may be enrolled as long as steroids are tapered off.
* Remission as defined by a CDAI ≤ 150.
* Women of childbearing potential, and men, must use medically acceptable methods of contraception [surgical sterilization, IUD, hormonal preparations, or double barrier method (e.g. condom or diaphragm, and spermicide)] throughout the study and for a period of 6 months after receiving the last injection.
* Screening lab results must be within prespecified limits: Hemoglobin ≥ 8.8 g/dl; SGOT/SGPT < 3 X the upper limit of normal; Neutrophil count ≥ 1.0 X 109/L & lymphocyte cont of ≥ 0.5 X 109/L
* Must have a documented PPD ≤ 5 mm, in patients taking steroids, within the month before randomization, or taking immunomodulators 2 months prior to randomization. Other patients must have documented PPD ≤ 10 mm prior to randomization. PPD must be preformed and documented by an appointed member of the investigatory stuff. Patients must have a normal chest radiograph (both posterior-anterior and lateral views), read by a certified radiologist, within 3 months prior to randomization.
* Commitment to adhere to study protocol requirements
* Negative stool cultures for enteric pathogens (Salmonella, Shigella, Campylobacter, Ova & parasites), and negative clostridium difficile toxin assay in stool.
* Patients are able to self-inject or have a designee or healthcare professional who can inject the study medication at the appropriate intervals.
* Patient's with long standing (>5Y), as well as recently diagnosed Crohn's disease ,will be eligible if they show radiologic (i.e. CT enterography, MR enterography , small bowel follow through) evidence, as well as laboratory (i.e. CRP, platelets level, fecal calprotectin, ESR ) evidence for an active inflammatory process within a 3 months period prior to the qualifying surgery

Exclusion Criteria:

* evidence of macroscopic inflammatory disease at the surgical margins or else ware, according to the surgeon
* Patients who discontinued anti TNF-alpha agents due to loss of efficacy or tolerability issues.
* Patients with temporary ileostomy.
* Patients with longstanding quiescent CD undergoing surgery for the treatment of a fibrostenotic lesion, without an active inflammatory disease process in the resected segment.
* Any of the following medications taken within 3 months prior to randomization: cyclosporine, tacrollimus, mycophenolate mofetil, or other investigational anti-inflammatory agents. Medication targeting the reduction of TNF-alpha (infliximab, golimumab, cetrolizumb pegol, etanercept), natalizumab, or other FDA approved biological agents may be administered up until to index surgery.
* Patient who have an ongoing active infection within the baseline period: intra-abdominal abscess, enteric infection as determined by stool cultures for bacteria, parasites and clostridium difficile toxin, other serious systemic bacterial infection within 3 months before randomization (e.g. Pneumonia; pyelonephritis; meningitis).
* Patients with active TB, patients in close contact to individuals with active TB, patients with latent TB whether receiving or not receiving prophylaxis.
* Patient that have or had an opportunistic infection within the last 6 months
* Patients seropositive to HIV, HBV, or HCV. Patients will be actively screened for HBV vaccination, and will be required to undergo vaccination according to international guidelines.
* Patients having current signs/symptoms of severe or progressive systemic disease: any progressive/uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or psychiatric illness.
* Patients after organ transplantation
* Any current or known malignancies
* Use of any investigational drug within 60 days prior to randomization
* Current/frequent use of NSAIDS (i.e. regular use of NSAIDS for more than 3 times a week for longer than 7 consecutive days during the trial period).
* Pregnant or lactating women
* Concomitant substance or alcohol abuse
* Subjects unable to self-inject or do not have a designee or healthcare professional who can inject the study medication.
* Subject unable to comply with the planned schedule of study visits and study procedures.
* Patients with short bowel syndrome
* Patients with previous small bowel surgeries

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with endoscopic recurrence at 12 months, as evaluated by the Rutgeerts endoscopic scoring system. | 52 weeks
  Primay outcome measure will assess the efficacy of adalimumab, compared to immunomodulator therapy in maintaining mucosal healing after 52 weeks (1 year).

SECONDARY OUTCOMES:
Proportion of patients in clinical remission at 12 months as assessed by the CDAI score. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erez F Scapa, M.D., Principal Investigator — Tel-Aviv Sourasky Medical Center, Affiliated to Tel-Aviv University; Iris Dotan, M.D., Study Director — Tel-Aviv Sourasky Medical Center, Affiliated to Tel-Aviv University
Locations (1):
- Department of Gastroenterology and Liver Diseases, Tel-Aviv Soursky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Regueiro M, Schraut W, Baidoo L, Kip KE, Sepulveda AR, Pesci M, Harrison J, Plevy SE. Infliximab prevents Crohn's disease recurrence after ileal resection. Gastroenterology. 2009 Feb;136(2):441-50.e1; quiz 716. doi: 10.1053/j.gastro.2008.10.051. Epub 2008 Oct 31. PMID 19109962
- [Derived] Hirsch A, Scapa E, Fliss-Isakov N, Tulchinsky H, Itzkowitz E, Kariv Y, Ron Y, Yanai H, White I, Yassin S, Cohen NA, Brazovski E, Dotan I, Maharshak N. Early Initiation of Adalimumab Significantly Diminishes Postoperative Crohn's Disease Endoscopic Recurrence and Is Superior to 6-Mercaptopurine Therapy: An Open-Label, Randomized Controlled Study. J Clin Med. 2023 Dec 10;12(24):7600. doi: 10.3390/jcm12247600. PMID 38137669